CLINICAL TRIAL: NCT02573181
Title: A Multicenter, Double-Blind Study of the Safety, Tolerability, and Immunogenicity of V114 Compared to Prevnar 13™ in Healthy Adults 65 Years of Age or Older Previously Vaccinated With 23-Valent Pneumococcal Polysaccharide Vaccine
Brief Title: Safety, Tolerability, and Immunogenicity of V114 Compared to Prevnar 13™ in PPSV23-vaccinated Healthy Adults ≥65 Years of Age (V114-007)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V114-007; V114-007 (Other: Merck Protocol Number)
Record Dates: First submitted 2015-10-08; First posted 2015-10-09 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- V114 (Experimental): Participants (≥65 years of age) who were vaccinated previously (≥1 year ago) with 23-valent pneumococcal polysaccharide vaccine will receive a single 0.5 mL intramuscular injection of V114 on Day 1.
  Interventions: Biological: V114
- Prevnar 13™ (Active Comparator): Participants (≥65 years of age) who were vaccinated previously (≥1 year ago) with 23-valent pneumococcal polysaccharide vaccine will receive a single 0.5 mL intramuscular injection of Prevnar 13™ on Day 1.
  Interventions: Biological: Prevnar 13™

INTERVENTIONS:
Biological: V114 — V114 contains 2 µg of serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F, and 4 μg of serotype 6B; and 30 µg of CRM₁₉₇ and 125 µg of Aluminum Phosphate Adjuvant (APA) per 0.5 mL dose.
  Arms: V114
Biological: Prevnar 13™ — Prevnar 13™ contains 2.2 μg of serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, and 23F, and 4.4 μg of serotype 6B; and 34 μg of CRM₁₉₇ and 125 μg of aluminum per 0.5mL dose.
  Arms: Prevnar 13™

SUMMARY:
This study is designed to assess the safety, tolerability, and immunogenicity of V114 compared with Prevnar 13™ in healthy adults 65 years of age or older previously vaccinated with 23-valent pneumococcal polysaccharide vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Is in good health (any underlying chronic illness must be documented to be in stable condition)
* Has documented proof of receipt of 23-valent pneumococcal polysaccharide vaccine ≥1 year prior to study entry
* Is a male or postmenopausal female

Exclusion Criteria:

* Has received prior administration of any pneumococcal vaccine other than 23-valent pneumococcal polysaccharide vaccine
* Has a history of invasive pneumococcal disease or known history of other culture-positive pneumococcal disease
* Has a known hypersensitivity to any component of the pneumococcal conjugate vaccine, or any diphtheria toxoid-containing vaccine
* Is known or suspected impairment of immune function
* Has received systemic corticosteroids for >=14 consecutive days and has not completed treatment <=30 days prior to study entry, or received systemic corticosteroids exceeding physiologic replacement doses within 14 days prior to study vaccination
* Has a coagulation disorder contraindicating intramuscular vaccination
* Receives immunosuppressive therapy, including chemotherapeutic agents used to treat cancer or other conditions, and treatments associated with organ or bone marrow transplantation, or autoimmune disease
* Has received a blood transfusion or blood products, including immunoglobulins within the 6 months before receipt of study vaccine or is scheduled to receive a blood transfusion or blood product within 30 days of receipt of study vaccine. Autologous blood transfusions are not considered an exclusion criterion
* Has participated in another clinical study of an investigational product within 2 months before the beginning of or any time during the duration of the current clinical study
* Is a user of recreational or illicit drugs or has had a recent history (within the last year) of drug or alcohol abuse or dependence.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 253 (Actual)
Dates: Start 2015-10-30 (Actual); Primary Completion 2016-01-28 (Actual); Study Completion 2016-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Peterson JT, Stacey HL, MacNair JE, Li J, Hartzel JS, Sterling TM, Benner P, Tamms GM, Musey LK. Safety and immunogenicity of 15-valent pneumococcal conjugate vaccine compared to 13-valent pneumococcal conjugate vaccine in adults >/=65 years of age previously vaccinated with 23-valent pneumococcal polysaccharide vaccine. Hum Vaccin Immunother. 2019;15(3):540-548. doi: 10.1080/21645515.2018.1532250. Epub 2018 Nov 14. PMID 30427749

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 17 study centers in the United States.
Groups:
- V114: Participants (≥65 years of age) who were vaccinated previously (≥1 year ago) with 23-valent pneumococcal polysaccharide vaccine received a single 0.5 mL intramuscular injection of V114 on Day 1.
- Prevnar 13™: Participants (≥65 years of age) who were vaccinated previously (≥1 year ago) with 23-valent pneumococcal polysaccharide vaccine received a single 0.5 mL intramuscular injection of Prevnar 13™ on Day 1.
Period: Overall Study
Arm/Group | V114 | Prevnar 13™
Started | 127 | 126
Vaccinated | 127 | 126
Completed | 127 | 126
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V114 | Prevnar 13™ | Total
Number analyzed (Participants) | 127 | 126 | 253
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.7 (5.8) | 72.7 (5.7) | 72.7 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 75 | 151
  Male | 51 | 51 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 19 | 39
  Not Hispanic or Latino | 107 | 107 | 214
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 8 | 15
  White | 120 | 118 | 238
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to Day 44 after vaccination
Population: All participants who received study vaccination are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 127 | 126
Percentage of Participants | 68.5 | 64.3
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Test type: Other — Difference in percentage with AEs; Difference = 4.2, 95% CI 2-sided [-7.4 to 15.8] — Difference and 95% CI calculated based on Miettinen & Nurminen method

2. Primary Outcome: Percentage of Participants With a Solicited Injection-site Adverse Event (AE)
Description: Solicited injection-site AEs consisted of erythema/redness, swelling, and pain/tenderness.
Time Frame: Up to Day 5 after vaccination
Population: All participants who received study vaccination are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 127 | 126
Percentage of Participants
  Erythema/Redness | 7.9 | 7.1
  Swelling | 14.2 | 6.3
  Tenderness/Pain | 55.1 | 44.4

3. Primary Outcome: Percentage of Participants With a Solicited Systemic Adverse Event (AE)
Description: Solicited systemic AEs consisted of fatigue, arthralgia, myalgia, and headache.
Time Frame: Up to Day 14 after vaccination
Population: All participants who received study vaccination are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 127 | 126
Percentage of Participants
  Fatigue | 18.1 | 19.0
  Arthralgia | 5.5 | 8.7
  Myalgia | 15.7 | 11.1
  Headache | 13.4 | 15.9
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Test type: Other — Difference in % with fatigue; Fatigue difference = -0.9, 95% CI 2-sided [-10.7 to 8.8] — Difference and 95% CI calculated based on the Miettinen & Nurminen method
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Test type: Other — Difference in % with arthralgia; Arthralgia difference = -3.2, 95% CI 2-sided [-10.2 to 3.4] — Difference and 95% CI calculated based on the Miettinen & Nurminen method
Statistical Analysis 3: Comparison: V114 vs Prevnar 13™; Test type: Other — Difference in % with myalgia; Myalgia difference = 4.6, 95% CI 2-sided [-3.9 to 13.3] — Difference and 95% CI calculated based on the Miettinen & Nurminen method
Statistical Analysis 4: Comparison: V114 vs Prevnar 13™; Test type: Other — Difference in % with headache; Headache difference = -2.5, 95% CI 2-sided [-11.4 to 6.4] — Difference and 95% CI calculated based on the Miettinen & Nurminen method

4. Primary Outcome: Geometric Mean Concentrations (GMCs) of Serotype-specific Immunoglobulin G (IgG)
Description: The IgG GMCs of each pneumococcal serotype were calculated on Day 1 (baseline) and Day 30 after vaccination. Concentrations were determined using pneumococcal electrochemiluminescence.
Time Frame: Baseline (Day 1) and Day 30 after vaccination
Population: Randomized and vaccinated participants with no protocol violations are included.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 127 | 126
µg/mL
  Serotype 1 Day 1: number analyzed (Participants) | 122 | 123
  Serotype 1 Day 1 | 1.11 [0.85 to 1.45] | 1.27 [.98 to 1.64]
  Serotype 1 Day 30: number analyzed (Participants) | 119 | 117
  Serotype 1 Day 30 | 3.31 [2.60 to 4.23] | 3.42 [2.61 to 4.47]
  Serotype 3 Day 1: number analyzed (Participants) | 122 | 123
  Serotype 3 Day 1 | 0.19 [0.15 to 0.23] | 0.19 [0.15 to 0.24]
  Serotype 3 Day 30: number analyzed (Participants) | 119 | 117
  Serotype 3 Day 30 | 0.72 [0.57 to 0.91] | 0.46 [0.36 to 0.58]
  Serotype 4 Day 1: number analyzed (Participants) | 122 | 123
  Serotype 4 Day 1 | 0.32 [0.25 to 0.41] | 0.33 [0.26 to 0.43]
  Serotype 4 Day 30: number analyzed (Participants) | 119 | 117
  Serotype 4 Day 30 | 1.13 [0.88 to 1.45] | 1.15 [0.88 to 1.51]
  Serotype 5 Day 1: number analyzed (Participants) | 122 | 123
  Serotype 5 Day 1 | 1.31 [1.01 to 1.70] | 1.48 [1.14 to 1.91]
  Serotype 5 Day 30: number analyzed (Participants) | 119 | 117
  Serotype 5 Day 30 | 2.69 [2.05 to 3.53] | 3.67 [2.75 to 4.90]
  Serotype 6A Day 1: number analyzed (Participants) | 122 | 123
  Serotype 6A Day 1 | 0.48 [0.36 to 0.64] | 0.47 [0.36 to 0.60]
  Serotype 6A Day 30: number analyzed (Participants) | 119 | 117
  Serotype 6A Day 30 | 3.85 [2.77 to 5.36] | 4.34 [3.17 to 5.94]
  Serotype 6B Day 1: number analyzed (Participants) | 122 | 123
  Serotype 6B Day 1 | 0.64 [0.48 to 0.87] | 0.67 [0.52 to 0.87]
  Serotype 6B Day 30: number analyzed (Participants) | 119 | 117
  Serotype 6B Day 30 | 3.74 [2.74 to 5.13] | 3.70 [2.72 to 5.04]
  Serotype 7F Day 1: number analyzed (Participants) | 122 | 123
  Serotype 7F Day 1 | 1.25 [0.94 to 1.67] | 1.01 [0.78 to 1.30]
  Serotype 7F Day 30: number analyzed (Participants) | 119 | 117
  Serotype 7F Day 30 | 3.85 [2.96 to 5.00] | 3.24 [2.54 to 4.12]
  Serotype 9V Day 1: number analyzed (Participants) | 122 | 123
  Serotype 9V Day 1 | 1.26 [0.99 to 1.61] | 1.04 [0.84 to 1.29]
  Serotype 9V Day 30: number analyzed (Participants) | 119 | 117
  Serotype 9V Day 30 | 3.79 [2.95 to 4.86] | 2.72 [2.17 to 3.41]
  Serotype 14 Day 1: number analyzed (Participants) | 122 | 123
  Serotype 14 Day 1 | 2.84 [2.12 to 3.81] | 4.10 [3.13 to 5.35]
  Serotype 14 Day 30: number analyzed (Participants) | 119 | 117
  Serotype 14 Day 30 | 5.46 [4.16 to 7.17] | 6.45 [5.00 to 8.32]
  Serotype 18C Day 1: number analyzed (Participants) | 122 | 123
  Serotype 18C Day 1 | 1.69 [1.28 to 2.22] | 1.76 [1.38 to 2.24]
  Serotype 18C Day 30: number analyzed (Participants) | 119 | 117
  Serotype 18C Day 30 | 6.85 [5.22 to 8.98] | 5.30 [4.15 to 6.77]
  Serotype 19A Day 1: number analyzed (Participants) | 122 | 123
  Serotype 19A Day 1 | 3.28 [2.54 to 4.24] | 3.29 [2.59 to 4.18]
  Serotype 19A Day 30: number analyzed (Participants) | 119 | 117
  Serotype 19A Day 30 | 9.3 [7.32 to 11.80] | 9.41 [7.76 to 11.41]
  Serotype 19F Day 1: number analyzed (Participants) | 122 | 123
  Serotype 19F Day 1 | 1.46 [1.10 to 1.94] | 1.45 [1.12 to 1.88]
  Serotype 19F Day 30: number analyzed (Participants) | 119 | 117
  Serotype 19F Day 30 | 5.06 [3.82 to 6.69] | 4.35 [3.35 to 5.66]
  Serotype 22F Day 1: number analyzed (Participants) | 122 | 123
  Serotype 22F Day 1 | 0.74 [0.57 to 0.96] | 0.68 [0.52 to 0.89]
  Serotype 22F Day 30: number analyzed (Participants) | 119 | 117
  Serotype 22F Day 30 | 2.57 [1.97 to 3.35] | 0.60 [0.46 to 0.79]
  Serotype 23F Day 1: number analyzed (Participants) | 122 | 123
  Serotype 23F Day 1 | 0.71 [0.54 to 0.93] | 0.73 [0.55 to 0.96]
  Serotype 23F Day 30: number analyzed (Participants) | 119 | 117
  Serotype 23F Day 30 | 4.01 [2.94 to 5.46] | 3.35 [2.41 to 4.65]
  Serotype 33F Day 1: number analyzed (Participants) | 122 | 123
  Serotype 33F Day 1 | 2.98 [2.24 to 3.96] | 3.30 [2.58 to 4.23]
  Serotype 33F Day 30: number analyzed (Participants) | 119 | 117
  Serotype 33F Day 30 | 6.57 [5.14 to 8.41] | 3.11 [2.40 to 4.04]

5. Primary Outcome: Geometric Mean Fold Rise (GMFR) From Baseline in Geometric Mean Concentrations (GMCs) of Serotype-specific Immunoglobulin G (IgG)
Description: The GMFR (Day 30 geometric mean concentration [GMC] / Day 1 GMC) from baseline (Day 1) to Day 30 of each pneumococcal IgG serotype was calculated. Concentrations of each pneumococcal serotype were determined using pneumococcal electrochemiluminescence.
Time Frame: Baseline (Day 1) and Day 30 after vaccination
Population: Randomized and vaccinated participants with no protocol violations, and with data for both Day 1 and Day 30, are included.
Measure: Geometric Mean (95% Confidence Interval); unit: GMFR
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 127 | 126
GMFR
  Serotype 1: number analyzed (Participants) | 119 | 117
  Serotype 1 | 2.98 [2.39 to 3.73] | 2.70 [2.17 to 3.35]
  Serotype 3: number analyzed (Participants) | 119 | 117
  Serotype 3 | 3.14 [2.54 to 3.88] | 2.03 [1.78 to 2.33]
  Serotype 4: number analyzed (Participants) | 119 | 117
  Serotype 4 | 3.37 [2.66 to 4.26] | 3.28 [2.73 to 3.95]
  Serotype 5: number analyzed (Participants) | 119 | 117
  Serotype 5 | 2.14 [1.82 to 2.50] | 2.39 [1.97 to 2.91]
  Serotype 6A: number analyzed (Participants) | 119 | 117
  Serotype 6A | 7.09 [5.71 to 8.79] | 8.24 [6.39 to 10.62]
  Serotype 6B: number analyzed (Participants) | 119 | 117
  Serotype 6B | 5.20 [4.19 to 6.46] | 4.92 [3.90 to 6.22]
  Serotype 7F: number analyzed (Participants) | 119 | 117
  Serotype 7F | 2.97 [2.44 to 3.63] | 3.03 [2.46 to 3.74]
  Serotype 9V: number analyzed (Participants) | 119 | 117
  Serotype 9V | 2.98 [2.42 to 3.67] | 2.57 [2.18 to 3.05]
  Serotype 14: number analyzed (Participants) | 119 | 117
  Serotype 14 | 1.90 [1.56 to 2.32] | 1.48 [1.28 to 1.72]
  Serotype 18C: number analyzed (Participants) | 119 | 117
  Serotype 18C | 4.06 [3.19 to 5.15] | 2.93 [2.37 to 3.64]
  Serotype 19A: number analyzed (Participants) | 119 | 117
  Serotype 19A | 2.85 [2.32 to 3.50] | 2.81 [2.35 to 3.37]
  Serotype 19F: number analyzed (Participants) | 119 | 117
  Serotype 19F | 3.37 [2.68 to 4.24] | 2.86 [2.36 to 3.46]
  Serotype 22F: number analyzed (Participants) | 119 | 117
  Serotype 22F | 3.27 [2.62 to 4.08] | 0.90 [0.87 to 0.94]
  Serotype 23F: number analyzed (Participants) | 119 | 117
  Serotype 23F | 5.26 [4.14 to 6.68] | 4.24 [3.34 to 5.38]
  Serotype 33F: number analyzed (Participants) | 119 | 117
  Serotype 33F | 2.22 [1.81 to 2.74] | 0.91 [0.88 to 0.95]

6. Primary Outcome: Percentage of Participants With ≥4-fold Rise From Baseline in Geometric Mean Concentrations (GMCs) of Serotype-specific Immunoglobulin G (IgG)
Description: The percentage of participants with ≥4-fold rise from baseline (Day 1) to Day 30 in GMCs of each pneumococcal serotype was calculated. Concentrations of each pneumococcal serotype were determined using pneumococcal electrochemiluminescence.
Time Frame: Baseline (Day 1) and Day 30 after vaccination
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 127 | 126
Percentage of Participants
  Serotype 1: number analyzed (Participants) | 119 | 117
  Serotype 1 | 32.8 [24.45 to 41.98] | 26.5 [18.77 to 35.45]
  Serotype 3: number analyzed (Participants) | 119 | 117
  Serotype 3 | 36.1 [27.53 to 45.45] | 17.1 [10.77 to 25.16]
  Serotype 4: number analyzed (Participants) | 119 | 117
  Serotype 4 | 36.1 [27.53 to 45.45] | 35.9 [27.24 to 45.29]
  Serotype 5: number analyzed (Participants) | 119 | 117
  Serotype 5 | 19.3 [12.66 to 27.58] | 23.9 [16.53 to 32.70]
  Serotype 6A: number analyzed (Participants) | 119 | 117
  Serotype 6A | 64.7 [55.42 to 73.24] | 65.0 [55.59 to 73.55]
  Serotype 6B: number analyzed (Participants) | 119 | 117
  Serotype 6B | 54.6 [45.24 to 63.77] | 46.2 [36.90 to 55.61]
  Serotype 7F: number analyzed (Participants) | 119 | 117
  Serotype 7F | 31.1 [22.93 to 40.23] | 33.3 [24.89 to 42.64]
  Serotype 9V: number analyzed (Participants) | 119 | 117
  Serotype 9V | 35.3 [26.76 to 44.58] | 23.9 [16.53 to 32.70]
  Serotype 14: number analyzed (Participants) | 119 | 117
  Serotype 14 | 18.5 [11.96 to 26.64] | 9.4 [4.79 to 16.20]
  Serotype 18C: number analyzed (Participants) | 119 | 117
  Serotype 18C | 46.2 [37.04 to 55.59] | 30.8 [22.57 to 39.97]
  Serotype 19A: number analyzed (Participants) | 119 | 117
  Serotype 19A | 31.1 [22.93 to 40.23] | 35.0 [26.45 to 44.41]
  Serotype 19F: number analyzed (Participants) | 119 | 117
  Serotype 19F | 35.3 [26.76 to 44.58] | 33.3 [24.89 to 42.64]
  Serotype 22F: number analyzed (Participants) | 119 | 117
  Serotype 22F | 31.9 [23.69 to 41.10] | 0.0 [0.0 to 3.10]
  Serotype 23F: number analyzed (Participants) | 119 | 117
  Serotype 23F | 52.9 [43.58 to 62.15] | 45.3 [36.08 to 54.77]
  Serotype 33F: number analyzed (Participants) | 119 | 117
  Serotype 33F | 24.4 [16.97 to 33.09] | 0.0 [0.0 to 3.10]

7. Secondary Outcome: Geometric Mean Titers (GMTs) of Serotype-specific Opsonophagocytic Killing Activity (OPA)
Description: The OPA GMTs of each pneumococcal serotype were calculated on Day 1 (baseline) and Day 30 after vaccination. Titer levels were determined with multiplexed OPA (MOPA-4).
Time Frame: Baseline (Day 1) and Day 30 after vaccination
Population: Randomized and vaccinated participants with no protocol violations are included.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 127 | 126
Titers
  Serotype 1 Day 1: number analyzed (Participants) | 122 | 120
  Serotype 1 Day 1 | 20.30 [14.87 to 27.70] | 24.24 [17.24 to 33.12]
  Serotype 1 Day 30: number analyzed (Participants) | 118 | 115
  Serotype 1 Day 30 | 109.25 [79.47 to 150.19] | 91.53 [65.77 to 127.37]
  Serotype 3 Day 1: number analyzed (Participants) | 122 | 119
  Serotype 3 Day 1 | 23.37 [17.56 to 31.09] | 26.71 [19.84 to 35.96]
  Serotype 3 Day 30: number analyzed (Participants) | 117 | 115
  Serotype 3 Day 30 | 145.24 [114.93 to 183.55] | 103.77 [81.94 to 131.41]
  Serotype 4 Day 1: number analyzed (Participants) | 122 | 120
  Serotype 4 Day 1 | 114.78 [76.28 to 172.72] | 96.28 [63.50 to 145.97]
  Serotype 4 Day 30: number analyzed (Participants) | 118 | 115
  Serotype 4 Day 30 | 881.94 [662.06 to 1174.84] | 924.82 [706.73 to 1210.21]
  Serotype 5 Day 1: number analyzed (Participants) | 122 | 120
  Serotype 5 Day 1 | 41.89 [28.38 to 61.83] | 39.52 [26.73 to 58.44]
  Serotype 5 Day 30: number analyzed (Participants) | 118 | 115
  Serotype 5 Day 30 | 183.10 [128.24 to 261.43] | 222.18 [154.84 to 318.81]
  Serotype 6A Day 1: number analyzed (Participants) | 121 | 120
  Serotype 6A Day 1 | 71.43 [44.92 to 113.61] | 46.57 [29.58 to 73.32]
  Serotype 6A Day 30: number analyzed (Participants) | 118 | 115
  Serotype 6A Day 30 | 2321.06 [1632.43 to 3300.19] | 2798.09 [2064.22 to 3792.87]
  Serotype 6B Day 1: number analyzed (Participants) | 122 | 120
  Serotype 6B Day 1 | 175.69 [113.53 to 271.90] | 132.41 [84.39 to 207.76]
  Serotype 6B Day 30: number analyzed (Participants) | 118 | 114
  Serotype 6B Day 30 | 2389.20 [1747.68 to 3266.19] | 2423.27 [1731.26 to 3391.90]
  Serotype 7F Day 1: number analyzed (Participants) | 122 | 119
  Serotype 7F Day 1 | 228.75 [150.65 to 347.35] | 205.76 [132.00 to 320.73]
  Serotype 7F Day 30: number analyzed (Participants) | 117 | 115
  Serotype 7F Day 30 | 1232.86 [905.89 to 1677.85] | 1664.85 [1328.78 to 2085.92]
  Serotype 9V Day 1: number analyzed (Participants) | 121 | 119
  Serotype 9V Day 1 | 320.81 [221.32 to 465.02] | 222.07 [146.84 to 335.85]
  Serotype 9V Day 30: number analyzed (Participants) | 118 | 115
  Serotype 9V Day 30 | 1962.51 [1450.32 to 2655.58] | 1387.45 [1008.48 to 1908.82]
  Serotype 14 Day 1: number analyzed (Participants) | 122 | 120
  Serotype 14 Day 1 | 451.24 [312.11 to 652.39] | 475.62 [349.01 to 648.15]
  Serotype 14 Day 30: number analyzed (Participants) | 118 | 115
  Serotype 14 Day 30 | 1228.80 [964.72 to 1565.18] | 899.66 [683.70 to 1183.84]
  Serotype 18C Day 1: number analyzed (Participants) | 122 | 120
  Serotype 18C Day 1 | 180.26 [121.60 to 267.21] | 205.56 [143.28 to 294.93]
  Serotype 18C Day 30: number analyzed (Participants) | 118 | 115
  Serotype 18C Day 30 | 1550.65 [1172.29 to 2051.13] | 1009.16 [728.59 to 1397.79]
  Serotype 19A Day 1: number analyzed (Participants) | 122 | 120
  Serotype 19A Day 1 | 498.71 [352.76 to 705.03] | 480.66 [348.91 to 662.17]
  Serotype 19A Day 30: number analyzed (Participants) | 118 | 115
  Serotype 19A Day 30 | 2078.60 [1650.03 to 2618.48] | 1861.84 [1480.24 to 2341.81]
  Serotype 19F Day 1: number analyzed (Participants) | 122 | 120
  Serotype 19F Day 1 | 145.50 [97.41 to 217.32] | 234.63 [168.86 to 362.02]
  Serotype 19F Day 30: number analyzed (Participants) | 117 | 115
  Serotype 19F Day 30 | 919.31 [690.56 to 1223.83] | 961.71 [747.20 to 1237.79]
  Serotype 22F Day 1: number analyzed (Participants) | 121 | 120
  Serotype 22F Day 1 | 173.09 [107.99 to 277.44] | 120.52 [73.92 to 196.49]
  Serotype 22F Day 30: number analyzed (Participants) | 118 | 114
  Serotype 22F Day 30 | 1761.25 [1255.38 to 2470.97] | 107.83 [64.66 to 179.80]
  Serotype 23F Day 1: number analyzed (Participants) | 122 | 120
  Serotype 23F Day 1 | 69.60 [47.54 to 101.91] | 48.74 [31.54 to 75.32]
  Serotype 23F Day 30: number analyzed (Participants) | 118 | 115
  Serotype 23F Day 30 | 846.33 [617.56 to 1159.85] | 572.82 [382.77 to 857.23]
  Serotype 33F Day 1: number analyzed (Participants) | 122 | 120
  Serotype 33F Day 1 | 1950.86 [1369.30 to 2779.43] | 2093.00 [1416.63 to 3092.30]
  Serotype 33F Day 30: number analyzed (Participants) | 118 | 113
  Serotype 33F Day 30 | 7856.78 [5750.01 to 10735.45] | 2572.78 [1800.33 to 3676.67]

8. Secondary Outcome: Geometric Mean Fold Rise (GMFR) From Baseline in Geometric Mean Titers (GMTs) of Serotype-specific Opsonophagocytic Killing Activity (OPA)
Description: The GMFR (Day 30 GMT / Day 1 GMT) from baseline (Day 1) to Day 30 of each OPA serotype was calculated. Titer levels were determined with multiplexed OPA (MOPA-4).
Time Frame: Baseline (Day 1) and Day 30 after vaccination
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: GMFR
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 127 | 126
GMFR
  Serotype 1: number analyzed (Participants) | 118 | 113
  Serotype 1 | 4.16 [3.09 to 5.58] | 3.33 [2.61 to 4.25]
  Serotype 3: number analyzed (Participants) | 117 | 112
  Serotype 3 | 5.06 [3.92 to 6.54] | 3.24 [2.61 to 4.02]
  Serotype 4: number analyzed (Participants) | 118 | 113
  Serotype 4 | 6.59 [4.52 to 9.60] | 7.94 [5.53 to 11.40]
  Serotype 5: number analyzed (Participants) | 118 | 113
  Serotype 5 | 3.94 [3.01 to 5.16] | 4.95 [3.65 to 6.71]
  Serotype 6A: number analyzed (Participants) | 117 | 113
  Serotype 6A | 25.19 [16.41 to 38.68] | 43.85 [27.28 to 70.49]
  Serotype 6B: number analyzed (Participants) | 118 | 112
  Serotype 6B | 11.83 [8.03 to 17.44] | 14.74 [9.85 to 22.07]
  Serotype 7F: number analyzed (Participants) | 117 | 112
  Serotype 7F | 4.77 [3.21 to 7.11] | 7.59 [5.03 to 11.44]
  Serotype 9V: number analyzed (Participants) | 117 | 112
  Serotype 9V | 5.79 [4.19 to 7.99] | 5.79 [4.10 to 8.17]
  Serotype 14: number analyzed (Participants) | 118 | 113
  Serotype 14 | 2.52 [1.86 to 3.42] | 1.89 [1.47 to 2.42]
  Serotype 18C: number analyzed (Participants) | 118 | 113
  Serotype 18C | 8.14 [5.80 to 11.42] | 4.93 [3.61 to 6.74]
  Serotype 19A: number analyzed (Participants) | 118 | 113
  Serotype 19A | 4.14 [3.10 to 5.53] | 3.83 [2.94 to 5.00]
  Serotype 19F: number analyzed (Participants) | 117 | 113
  Serotype 19F | 5.55 [3.98 to 7.74] | 4.02 [3.11 to 5.19]
  Serotype 22F: number analyzed (Participants) | 117 | 112
  Serotype 22F | 8.88 [5.44 to 14.48] | 0.85 [0.61 to 1.19]
  Serotype 23F: number analyzed (Participants) | 118 | 113
  Serotype 23F | 10.41 [7.18 to 15.10] | 9.58 [6.47 to 14.19]
  Serotype 33F: number analyzed (Participants) | 118 | 112
  Serotype 33F | 3.91 [2.76 to 5.54] | 1.03 [0.88 to 1.20]

9. Secondary Outcome: Percentage of Participants With ≥4-fold Rise From Baseline in Geometric Mean Titers (GMTs) of Serotype-specific Opsonophagocytic Killing Activity (OPA)
Description: The percentage of participants with ≥4-fold rise from baseline (Day 1) to Day 30 in GMTs of each pneumococcal serotype was calculated. Titer levels were determined with multiplexed OPA (MOPA-4).
Time Frame: Baseline (Day 1) and Day 30 after vaccination
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 127 | 126
Percentage of Participants
  Serotype 1: number analyzed (Participants) | 118 | 113
  Serotype 1 | 40.7 [31.73 to 50.11] | 33.6 [25.01 to 43.12]
  Serotype 3: number analyzed (Participants) | 117 | 112
  Serotype 3 | 53.8 [44.39 to 63.10] | 39.3 [30.19 to 48.96]
  Serotype 4: number analyzed (Participants) | 118 | 113
  Serotype 4 | 44.1 [34.94 to 53.50] | 54.9 [45.23 to 64.25]
  Serotype 5: number analyzed (Participants) | 118 | 113
  Serotype 5 | 44.9 [35.75 to 54.34] | 50.4 [40.88 to 59.98]
  Serotype 6A: number analyzed (Participants) | 117 | 113
  Serotype 6A | 71.8 [62.73 to 79.72] | 77.0 [68.13 to 84.39]
  Serotype 6B: number analyzed (Participants) | 118 | 112
  Serotype 6B | 62.7 [53.33 to 71.44] | 67.0 [57.44 to 75.56]
  Serotype 7F: number analyzed (Participants) | 117 | 112
  Serotype 7F | 41.0 [32.02 to 50.50] | 50.0 [40.40 to 59.60]
  Serotype 9V: number analyzed (Participants) | 117 | 112
  Serotype 9V | 47.9 [38.54 to 57.29] | 44.6 [35.24 to 54.33]
  Serotype 14: number analyzed (Participants) | 118 | 113
  Serotype 14 | 18.6 [12.07 to 26.86] | 15.9 [9.72 to 24.00]
  Serotype 18C: number analyzed (Participants) | 118 | 113
  Serotype 18C | 54.2 [44.82 to 63.44] | 43.4 [34.07 to 53.01]
  Serotype 19A: number analyzed (Participants) | 118 | 113
  Serotype 19A | 37.3 [28.56 to 46.67] | 37.2 [28.26 to 46.76]
  Serotype 19F: number analyzed (Participants) | 117 | 113
  Serotype 19F | 40.2 [31.22 to 49.64] | 38.1 [29.08 to 47.67]
  Serotype 22F: number analyzed (Participants) | 117 | 112
  Serotype 22F | 50.4 [41.03 to 59.80] | 9.8 [5.01 to 16.89]
  Serotype 23F: number analyzed (Participants) | 118 | 113
  Serotype 23F | 61.0 [51.61 to 69.86] | 52.2 [42.61 to 61.70]
  Serotype 33F: number analyzed (Participants) | 118 | 112
  Serotype 33F | 38.1 [29.35 to 47.53] | 6.3 [2.55 to 12.45]

ADVERSE EVENTS:
Time Frame: Nonserious AEs were monitored for up to 14 days after vaccination. Deaths and serious AEs (SAEs) were monitored up to 30 days after vaccination.
Description: All participants who received study vaccination are included in the safety analysis.
Groups:
- Prevnar 13®: Participants (≥65 years of age) who were vaccinated previously (≥1 year ago) with 23-valent pneumococcal polysaccharide vaccine received a single 0.5 mL intramuscular injection of Prevnar 13™ on Day 1.
Arm/Group | V114 | Prevnar 13®
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/126
Serious Adverse Events (participants affected / at risk) | 0/127 | 2/126
Other Adverse Events (participants affected / at risk) | 86/127 | 74/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=127) | Prevnar 13® (N=126)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=127) | Prevnar 13® (N=126)
Fatigue (General disorders) | 23 (27) | 24 (30)
Injection site erythema (General disorders) | 12 (12) | 10 (10)
Injection site pain (General disorders) | 73 (78) | 58 (61)
Injection site swelling (General disorders) | 20 (21) | 8 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 11 (15)
Myalgia (Musculoskeletal and connective tissue disorders) | 20 (23) | 14 (15)
Headache (Nervous system disorders) | 17 (20) | 20 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.